CLINICAL TRIAL: NCT01477424
Title: A Single-centre, Open-label, Three-period Study of the Pharmacokinetic Effect of PA21 on Warfarin in Healthy Male and Female Adults
Brief Title: A Drug-Drug Interaction Study of Warfarin and PA21
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PA-DDI-005
Record Dates: First submitted 2011-11-16; First posted 2011-11-22 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Drug Interaction Potentiation
Keywords: Drug-drug interaction; Pharmacokinetics; PA21
MeSH Terms: interventions — Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PA21 and Warfarin with food (Experimental): The maximum dose of PA21 will be 15.0 g/day. The maximum dose of Warfarin will be 10 mg/day
  Interventions: Drug: PA21; Drug: Warfarin
- No PA21; Warfarin with food (Experimental): The maximum dosage of Warfarin will be 10 mg/day
  Interventions: Drug: Warfarin
- PA21 with food and Warfarin 2hrs later (Experimental): The maximum dose of PA21 will be 15 g/day. The maximum dose of Warfarin will be 10 mg/day
  Interventions: Drug: PA21; Drug: Warfarin

INTERVENTIONS:
Drug: PA21 — The maximum dose of PA21 will be 15.0 g/day.
  Arms: PA21 and Warfarin with food; PA21 with food and Warfarin 2hrs later
Drug: Warfarin — The maximum dosage of Warfarin will be 10 mg/day

SUMMARY:
The purpose of this study is to determine if Warfarin is affected by PA21.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Written informed consent

Exclusion Criteria:

* No significant medical conditions
* Pregnancy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from time zero to 24 hours (AUC0-24) | pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post Warfarin dose on Days 0, 11, 22
  Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours
Area Under the Curve from time zero to infinite (AUC0-infinity) | pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120, 144 and 168 hours post Warfarin dose on Days 0, 11, 22
  Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time
Maximum observed plasma concentration (Cmax) | pre-dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 120 and 168 hours post Warfarin dose on days 0, 11, 22

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K Willsie, MD, Principal Investigator — PRA International - Clinical Pharmacology Center
Locations (1):
- PRA International - Clinical Pharmacology Center, Lenexa, Kansas, United States